CLINICAL TRIAL: NCT04505644
Title: Is Lidocaine Patch as Effective as Intravenous Lidocaine in Pain and Illus Reduction After Cesarean Section? A Randomized Clinical Trial
Brief Title: Lidocaine Patch Versus Intravenous Lidocaine in Pain Relief After Cesarean Section
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, hany farouk, A Professor, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: aswu/279/6/18
Record Dates: First submitted 2020-08-06; First posted 2020-08-10 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Cesarean Section Complications
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Intervention Model Description: double blind randomized controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blind randomized controlled study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- lidocaine patch (Experimental): 5% lidocaine patch applied at 12 hours after cesarean delivery and removed 24 hours after delivery. A second 5% lidocaine patch applied at 36 hours after cesarean delivery and removed at 48 hours after delivery.
  Interventions: Drug: lidocaine patch
- IV lidocaine (Active Comparator): received i.v. lidocaine infusion after induction of anesthesia, 2 mg/min if body weight >70 kg or 1 mg/min if body weight <70 kg.
  Interventions: Drug: IV lidocaine
- IV saline infusion +Sham patch (Placebo Comparator): received i.v. saline infusion +Sham patch containing no study medication applied at 12 hours after cesarean delivery and removed 24 hours after delivery. A second sham patch containing no study medication applied at 36 hours after cesarean delivery and removed at 48 hours after delivery.
  Interventions: Drug: IV saline infusion +Sham patch

INTERVENTIONS:
Drug: lidocaine patch — Sham patch containing no study medication applied at 12 hours after cesarean delivery and removed 24 hours after delivery. A second sham patch containing no study medication applied at 36 hours after cesarean delivery and removed at 48 hours after delivery.
  Other Names: ;lidocaine patch
  Arms: lidocaine patch
Drug: IV lidocaine — received i.v. lidocaine infusion after induction of anesthesia, 2 mg/min if body weight >70 kg or 1 mg/min if body weight <70 kg.
  Arms: IV lidocaine
Drug: IV saline infusion +Sham patch — received i.v. saline infusion +Sham patch containing no study medication applied at 12 hours after cesarean delivery and removed 24 hours after delivery. A second sham patch containing no study medication applied at 36 hours after cesarean delivery and removed at 48 hours after delivery.
  Other Names: placebo
  Arms: IV saline infusion +Sham patch

SUMMARY:
To evaluate the efficacy of lidocaine patch applied around wound in reduction of postoperative pain and illus compared to intravenous lidocaine infusion and placebo after cesarean section.

DETAILED DESCRIPTION:
The use of lidocaine as a local anesthetic is a common and widely used in practice. Lidocaine patches can be used for localized pain control and can be placed every 24 hours. The use of lidocaine patches in post-operative patients has been reported in one case report in obstetric literature. There is one study that reports decreased immediate postoperative pain when lidocaine patches were placed at laparoscopic port sites following gynecologic surgery as measured by visual analog scale score and the Prince Henry and 5-point verbal rating pain scale . There have been no studies looking at the impact of lidocaine patches in obstetric surgical procedures, specifically cesarean sections.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Primary or secondary cesarean delivery
* Able to consent to research study

Exclusion Criteria:

* 3 or more prior cesarean deliveries
* History of abdominoplasty
* History of abdominal hernia repair with mesh
* Allergy to lidocaine
* Allergy to adhesives in medical tape
* Women who received general anesthesia for their cesarean delivery
* Women with active substance abuse
* Women methadone or suboxone for a history of opiate abuse

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Patients need to be pregnant and undergoing a cesarean delivery
Enrollment: 180 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2021-03-30 (Estimated); Study Completion 2021-05-30 (Estimated)

PRIMARY OUTCOMES:
Total dose of opioids received in the first 24 hours following Cesarean | 24 hours
  The total dose of opioids received in the first 24 hours following Cesarean delivery measured as oral morphine equivalents. This total dose will be calculated for every subject in the study, and the average and standard deviation (or appropriate non-parametric values if the data is not normally distributed) will be compared between the subjects randomized to the intervention arm and the placebo arm of the study.
Post-operative pain score at 24 hours post-operatively | 24 hours
  Assessment of pain using visual analog scale 0-10, 0 = minimum and 10 = maximum scores

SECONDARY OUTCOMES:
Incidence of complications of lidocaine use | 72 hours
  Complications of lidocaine use include local burning, nausea, dizziness, drowsiness, serious skin reactions such as blistering, confusion, blurred vision, ringing in the ears, and allergies and hypersensitivities.
  Definition: Patient reported side effects which will be reported as frequencies of occurrence
Return of bowel function | 72 hours
  Return of bowel function (measured in hours from completion of surgery to passage of flatus) Measured in hours from completion of surgery to passage of flatus. This will be reported as a continuous variable for the number of hours following surgery to flatus

CONTACTS AND LOCATIONS:
Overall Officials: nahla w Shady, md, Study Chair — Aswan universirty
Locations (1):
- Aswan University Hospital, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: No